CLINICAL TRIAL: NCT06766006
Title: A Multicentric Left Ventricular Venting Strategy Comparison in Patients Receiving Venoarterial Extracorporeal Life Support
Brief Title: ECMO LEft Ventricle UNloading Strategy
Acronym: ECMOLENS
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0112
Record Dates: First submitted 2023-12-14; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Shock, Cardiogenic; Cardiac Arrest; Extracorporeal Membrane Oxygenation Complication
Keywords: Extracorporeal Membrane Oxygenation; Left ventricle unloading; Cardiogenic shock; Cardiac Arrest; Mechanical Circulatory Supports
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest | interventions — Drug Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VA ECLS patients: All patients undergoing VA ECLS will be enrolled. Patients without VA ECLS will not be considered. Centers will follow their standard protocols for the management of patients on VA ECLS.
  Interventions: Procedure: Venoarterial extracorporeal life support (VA ECLS) implant

INTERVENTIONS:
Procedure: Venoarterial extracorporeal life support (VA ECLS) implant — Implantation of venoarterial extracorporeal life support implant for refractory cardiogenic shock or cardiac arrest of any cause.

SUMMARY:
The present study is an International multicentric prospective observational cohort study. This will be an international research campaign to prospectively collect and analyze clinical data of all VA ECLS patients admitted to participating ICUs with a focus on LV venting modalities. The aims of the study are:

* To investigate the meaning of LV overload during veno-arterial (VA) extracorporeal life support;
* To extensively describe the left ventricular (LV) unloading strategy during VA extracorporeal life support in a large prospective international cohort.
* To compare different strategies to unload the left ventricular in terms of efficacy and outcomes;

DETAILED DESCRIPTION:
Cardiogenic shock and cardiac arrest are among the most lethal manifestations of acute cardiovascular disease, both burdened by extremely high in-hospital mortality rates. Extracorporeal life support is increasingly used either in adults or children with acutely impaired cardiac function refractory to conventional medical management, mainly in profound cardiogenic shock and refractory cardiac arrest. Veno-arterial extracorporeal life support works as a partial cardiopulmonary bypass draining the venous circulation directly into the systemic circulation. Veno-arterial extracorporeal life support provides biventricular support and provides respiratory gas exchange. One of the most important issues occurring during veno-arterial extracorporeal life support is the effect of the retrograde aortic flow which causes a marked increase in the left ventricular afterload with detrimental effects on myocardial performance. Left ventricular overload increases wall stress and myocardial oxygen consumption, jeopardizing ventricular recovery. Nowadays, different techniques are available for unloading the left chambers. However, despite the increasing worldwide experience with extracorporeal life support and the increased knowledge on the benefits of left ventricular unloading, the best veno-arterial extracorporeal life support configuration to achieve hemodynamic support, myocardial recovery, and left ventricular unloading, is still a matter of debate.

This is a prospective clinical study which is observational. The aims of the study are:

* To extensively describe the left ventricular unloading strategy during veno-arterial extracorporeal life support in a large prospective international cohort, providing detailed information on indications, timing, type and modality among a wide spectrum of clinical conditions
* To compare different strategies to unload the left ventricular in terms of efficacy and outcomes
* To provide a common definition of left ventricular overload by collecting clinical, hemodynamic data and radiological information before and after unloading.

Demographics, clinical, instrumental and laboratory data prior and post implantation of veno-arterial extracorporeal life support will be collected. No interventions on top on the ones necessary as a standard of care will be taken.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing VA ECLS will be enrolled.

Exclusion Criteria:

* Patients without VA ECMO will not be considered

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by cardiogenic shock or cardiac arrest independent of etiology supported with VA ECLS.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Day 30
  Death during hospital stay
Overload detection, Echocardiographic parameters | Within 12 hours before the applied unloading technique
  Presence of left ventricle (LV) overload (defined as: aortic valve opening impairment and/or smoke like effect and/or LA distension and/or LV distension).
  The aforementioned criteria are defined as follows:
  * Aortic valve opening impairment: Aortic valve does not open every beat.
  * Smoke like effect: spontaneous echo contrast inside left ventricle chamber.
  * Left Atrium (LA) distension: male/female LA volume/body surface area (BSA)>=34 or increase>15%
  * LV distension: LV end-diastolic volume (ml) >150 ml, male; female LV end-diastolic volume (ml) >106 ml or increase>15%
Unloading effectiveness, Echocardiographic parameters | 12 hours after the unloading technique implementation
  Echocardiographic qualitative parameters:
  * aortic valve opening (yes/no)
  * smoke like effect (yes/no)
  * LA distension (yes/no)
  * LV distension (yes/no)
  * inferior vena cava collapse/dilation (yes/no)
  * grade of mitral regurgitation (mild/moderatre/severe)
  Echocardiographic quantitative parameters:
  * LV end-diastolic diameter (mm)
  * LV end-diastolicvolume (ml)
  * LV end-systolic diameter (mm)
  * LV end-systolic volume(ml)
  * LA volume (ml)
  * E/E' septal and lateral (ratio, no unit of measurement )
  * systolic pulmonary artery pressure (mmHg)

SECONDARY OUTCOMES:
Unloading Effectiveness, Qualitative echocardiographic parameters | 12 hours after the unloading technique implementation
  Unloading effectiveness, qualitative evaluation (yes/no) ( any of the following criteria: restored aortic valve opening (yes/no) and/or solved smoke like effect (yes/no) and/or reduced LA distension (yes/no) and/or reduced LV distension (yes/no) and/or decreased grade of mitral regurgitation)
Major adverse events | Day 30
  Cerebral injury (stroke, transitory ischemic attack, intracranial hemorrhage and seizures by electroencephalogram), acute kidney injury requiring continuous renal replacement therapy, hemolysis (defined as increased free hemoglobin level, peripheral vascular damage, infections (defined as positive bacterial, fungal or viral culture or polymerase chain reaction test), coagulation disorders (either thrombosis or hemorrhage) and ECLS failure (pump or oxygenator failure, or both), liver and kidney organ function.
Left Ventricular functional status | Day 30
  Left ventricle Ejection fraction (%)
LVAD Implementation | Day 30
  LVAD implant
Heart transplant | Day 30
  Heart transplant
Neurological status at discharge | Day 30
  Cerebral Performance Category (CPC)

OTHER OUTCOMES:
Unloading Effectiveness, Quantitative echocardiographic parameters, LV end-diastolic diameter (mm) | 12 hours after the unloading technique implementation
  LV end-diastolic diameter (mm)
Unloading Effectiveness, Quantitative echocardiographic parameters, LV end-diastolic volume (ml) | 12 hours after the unloading technique implementation
  LV end-diastolic volume (ml)
Unloading Effectiveness, Quantitative echocardiographic parameters, LV end-systolic diameter (mm) | 12 hours after the unloading technique implementation
  LV end-systolic diameter (mm)
Unloading Effectiveness, Quantitative echocardiographic parameters, LV end-systolic volume(ml) | 12 hours after the unloading technique implementation
  LV end-systolic volume(ml)
Unloading Effectiveness, Quantitative echocardiographic parameters, LA volume (ml) | 12 hours after the unloading technique implementation
  LA volume (ml)
Unloading Effectiveness, Quantitative echocardiographic parameters, E/E' septal and lateral (ratio, no unit of measurement ) | 12 hours after the unloading technique implementation
  E/E' septal and lateral (ratio, no unit of measurement )
Unloading Effectiveness, Quantitative echocardiographic parameters, Systolic pulmonary artery pressure (mmHg) | 12 hours after the unloading technique implementation
  Systolic pulmonary artery pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Camboni D, Schmid C. To vent or not on veno-arterial extracorporeal membrane oxygenation, does it improve myocardial recovery and outcome? J Thorac Dis. 2017 Dec;9(12):4915-4918. doi: 10.21037/jtd.2017.11.98. No abstract available. PMID 29312691
- [Background] Schrage B, Becher PM, Bernhardt A, Bezerra H, Blankenberg S, Brunner S, Colson P, Cudemus Deseda G, Dabboura S, Eckner D, Eden M, Eitel I, Frank D, Frey N, Funamoto M, Gossling A, Graf T, Hagl C, Kirchhof P, Kupka D, Landmesser U, Lipinski J, Lopes M, Majunke N, Maniuc O, McGrath D, Mobius-Winkler S, Morrow DA, Mourad M, Noel C, Nordbeck P, Orban M, Pappalardo F, Patel SM, Pauschinger M, Pazzanese V, Reichenspurner H, Sandri M, Schulze PC, H G Schwinger R, Sinning JM, Aksoy A, Skurk C, Szczanowicz L, Thiele H, Tietz F, Varshney A, Wechsler L, Westermann D. Left Ventricular Unloading Is Associated With Lower Mortality in Patients With Cardiogenic Shock Treated With Venoarterial Extracorporeal Membrane Oxygenation: Results From an International, Multicenter Cohort Study. Circulation. 2020 Dec;142(22):2095-2106. doi: 10.1161/CIRCULATIONAHA.120.048792. Epub 2020 Oct 9. PMID 33032450
- [Background] Haneya A, Philipp A, Diez C, Schopka S, Bein T, Zimmermann M, Lubnow M, Luchner A, Agha A, Hilker M, Hirt S, Schmid C, Muller T. A 5-year experience with cardiopulmonary resuscitation using extracorporeal life support in non-postcardiotomy patients with cardiac arrest. Resuscitation. 2012 Nov;83(11):1331-7. doi: 10.1016/j.resuscitation.2012.07.009. Epub 2012 Jul 20. PMID 22819880
- [Background] Arlt M, Philipp A, Voelkel S, Schopka S, Husser O, Hengstenberg C, Schmid C, Hilker M. Early experiences with miniaturized extracorporeal life-support in the catheterization laboratory. Eur J Cardiothorac Surg. 2012 Nov;42(5):858-63. doi: 10.1093/ejcts/ezs176. Epub 2012 May 3. PMID 22555310
- [Background] Donker DW, Brodie D, Henriques JPS, Broome M. Left ventricular unloading during veno-arterial ECMO: a review of percutaneous and surgical unloading interventions. Perfusion. 2019 Mar;34(2):98-105. doi: 10.1177/0267659118794112. Epub 2018 Aug 16. PMID 30112975
- [Background] Meani P, Lorusso R, Pappalardo F. ECPella: Concept, Physiology and Clinical Applications. J Cardiothorac Vasc Anesth. 2022 Feb;36(2):557-566. doi: 10.1053/j.jvca.2021.01.056. Epub 2021 Feb 6. PMID 33642170
- [Background] Meani P, Gelsomino S, Natour E, Johnson DM, Rocca HB, Pappalardo F, Bidar E, Makhoul M, Raffa G, Heuts S, Lozekoot P, Kats S, Sluijpers N, Schreurs R, Delnoij T, Montalti A, Sels JW, van de Poll M, Roekaerts P, Poels T, Korver E, Babar Z, Maessen J, Lorusso R. Modalities and Effects of Left Ventricle Unloading on Extracorporeal Life support: a Review of the Current Literature. Eur J Heart Fail. 2017 May;19 Suppl 2:84-91. doi: 10.1002/ejhf.850. PMID 28470925
- [Background] Meani P, Delnoij T, Raffa GM, Morici N, Viola G, Sacco A, Oliva F, Heuts S, Sels JW, Driessen R, Roekaerts P, Gilbers M, Bidar E, Schreurs R, Natour E, Veenstra L, Kats S, Maessen J, Lorusso R. Protracted aortic valve closure during peripheral veno-arterial extracorporeal life support: is intra-aortic balloon pump an effective solution? Perfusion. 2019 Jan;34(1):35-41. doi: 10.1177/0267659118787426. Epub 2018 Jul 19. PMID 30024298
- [Background] Patel SM, Lipinski J, Al-Kindi SG, Patel T, Saric P, Li J, Nadeem F, Ladas T, Alaiti A, Phillips A, Medalion B, Deo S, Elgudin Y, Costa MA, Osman MN, Attizzani GF, Oliveira GH, Sareyyupoglu B, Bezerra HG. Simultaneous Venoarterial Extracorporeal Membrane Oxygenation and Percutaneous Left Ventricular Decompression Therapy with Impella Is Associated with Improved Outcomes in Refractory Cardiogenic Shock. ASAIO J. 2019 Jan;65(1):21-28. doi: 10.1097/MAT.0000000000000767. PMID 29489461
- [Background] Grandin EW, Nunez JI, Willar B, Kennedy K, Rycus P, Tonna JE, Kapur NK, Shaefi S, Garan AR. Mechanical Left Ventricular Unloading in Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation. J Am Coll Cardiol. 2022 Apr 5;79(13):1239-1250. doi: 10.1016/j.jacc.2022.01.032. PMID 35361346
- [Background] Raffa GM, Kowalewski M, Meani P, Follis F, Martucci G, Arcadipane A, Pilato M, Maessen J, Lorusso R; ECMO in TAVI Investigators Group (ETIG). In-hospital outcomes after emergency or prophylactic veno-arterial extracorporeal membrane oxygenation during transcatheter aortic valve implantation: a comprehensive review of the literature. Perfusion. 2019 Jul;34(5):354-363. doi: 10.1177/0267659118816555. Epub 2019 Jan 11. PMID 30632894
- [Background] Pappalardo F, Schulte C, Pieri M, Schrage B, Contri R, Soeffker G, Greco T, Lembo R, Mullerleile K, Colombo A, Sydow K, De Bonis M, Wagner F, Reichenspurner H, Blankenberg S, Zangrillo A, Westermann D. Concomitant implantation of Impella(R) on top of veno-arterial extracorporeal membrane oxygenation may improve survival of patients with cardiogenic shock. Eur J Heart Fail. 2017 Mar;19(3):404-412. doi: 10.1002/ejhf.668. Epub 2016 Oct 6. PMID 27709750